CLINICAL TRIAL: NCT01130688
Title: Phase I Study to Evaluate the Safety of Zileuton (Zyflo) in Combination With Imatinib Mesylate (Gleevec) in Patients With Chronic Myelogenous Leukemia
Brief Title: Safety of Zileuton (Zyflo) in Combination With Imatinib Mesylate (Gleevec) in CML.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Jan Cerny, Principal Investigator, University of Massachusetts, Worcester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UM200905
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2013-01

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: Leukemia; Zileuton; myeloproliferative neoplasm
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia; Myeloproliferative Disorders | interventions — zileuton

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm of experimental drug combination (Experimental)
  Interventions: Drug: Zileuton

INTERVENTIONS:
Drug: Zileuton — Imatinib combined with Zileuton
  Other Names: Zyflo

SUMMARY:
The leukemic stem cells (LSCs) are cells that self- renew and give rise to leukemia. Eradication of LSC is required for cure. In chronic myelogenous leukemia (CML) LSCs are not eradicated by imatinib (Gleevec) alone. Recent discovery by Dr. Shaoguang Li at University of Massachusetts indicates that the LSCs can be targeted by a new drug zileuton (Chen et al. Nature Genetics 2009; 41:783-792). Zileuton (approved for asthma) will be tested in a combination with Gleevec. This combination has not been used previously to treat leukemia.

This is a Phase I study. The goal of this research is to evaluate the safety of the standard anti-cancer drug imatinib and experimental drug zileuton.

DETAILED DESCRIPTION:
More than twenty two thousand people live with chronic myelogenous leukemia in the United States and more than five thousand people are expected to be diagnosed this year. The majority of patients with this disease are diagnosed in what is called the chronic phase. The standard treatment for this phase of the disease is therapy with a medication called imatinib. This treatment can diminish the amount of disease to very low levels that only very sensitive and specialized techniques can measure; it does not, however, provide a cure.

Dr. Shaoguang Li and colleagues at University of Massachusetts have published a unique discovery that the arachidonate 5-lipoxygenase (5-LO) gene (Alox5) is a critical regulator for LSCs in BCR-ABL-induced CML (Chen Y et al. Loss of the Alox5 gene impairs leukemia stem cells and prevents chronic myeloid leukemia. Nature Genetics 41:783-792, 2009). In the absence of Alox5, BCR-ABL failed to induce CML in preclinical studies. While deficiency in Alox5 had no effect on normal hematopoiesis, impairment of the LSCs function through differentiation and cell division of CML LSCs was observed. This defect led to a depletion of LSCs and a failure of CML development. Treatment with a 5-LO inhibitor (zileuton) also impaired the function of LSCs and prolonged survival. These results demonstrate that a specific target gene can be found in cancer stem cells and its inhibition can completely inhibit the function of these stem cells. These findings provide an exciting opportunity to develop the first anti-cancer stem cell therapy for treating CML.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CML in chronic phase (patients already on imatinib)
* Presence of Philadelphia chromosome or bcr-abl rearrangement
* Age ≥ 18 years
* ECOG performance status ≤ 2
* Written informed consent

Exclusion Criteria:

* Hepatic dysfunction (serum bilirubin ≥ 2 x ULN, and/or ALT ≥ 3 x ULN, and/or AST ≥ 3 x ULN)
* Renal dysfunction (creatinine ≥ 200 μmol/l or 2.3 mg/dl)
* Severe cardiac dysfunction (NYHA classification III-IV)
* Severe pulmonary or neurologic disease
* Pregnant or lactating females
* Patients with a history of active malignancy during the past 5 years with the exception of nonmetastatic skin cancer (e.g. treated squamous or basal cell carcinoma) or stage 0 cervical carcinoma
* Patients known to be HIV-positive
* Patients with active, uncontrolled infections
* Male and female patients of reproductive potential who are not practicing effective means of contraception
* Patients with known allergic reaction or intolerance to either imatinib or zileuton
* Patients requiring anticoagulation therapy with coumadin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-01; Primary Completion 2012-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To define toxicity and safety profile of zileuton combined with imatinib in patients with CML | Throughout the study

SECONDARY OUTCOMES:
To assess the efficacy of zileuton combined with imatinib in terms of (See Description) | Throughout the study
  * Level of 5-lipoxygenase (5-LO) blockade
  * The rate of complete hematological response
  * The rate of complete cytogenetic response
  * The rate of major molecular response

CONTACTS AND LOCATIONS:
Overall Officials: Jan Cerny, MD, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

REFERENCES:
- [Result] Chen Y, Hu Y, Zhang H, Peng C, Li S. Loss of the Alox5 gene impairs leukemia stem cells and prevents chronic myeloid leukemia. Nat Genet. 2009 Jul;41(7):783-92. doi: 10.1038/ng.389. Epub 2009 Jun 7. PMID 19503090
- [Result] Druker BJ, Guilhot F, O'Brien SG, Gathmann I, Kantarjian H, Gattermann N, Deininger MW, Silver RT, Goldman JM, Stone RM, Cervantes F, Hochhaus A, Powell BL, Gabrilove JL, Rousselot P, Reiffers J, Cornelissen JJ, Hughes T, Agis H, Fischer T, Verhoef G, Shepherd J, Saglio G, Gratwohl A, Nielsen JL, Radich JP, Simonsson B, Taylor K, Baccarani M, So C, Letvak L, Larson RA; IRIS Investigators. Five-year follow-up of patients receiving imatinib for chronic myeloid leukemia. N Engl J Med. 2006 Dec 7;355(23):2408-17. doi: 10.1056/NEJMoa062867. PMID 17151364